CLINICAL TRIAL: NCT01848158
Title: Safety, Feasibility & Effectiveness of Acupuncture as an Adjunct to Pharmacologic Treatment for Sedation and Analgesia in Mechanically Ventilated PICU Patients - A Pilot Study
Brief Title: Acupuncture to Improve Comfort of Children on a Ventilator in the Intensive Care Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Lin Di Gennaro, Jane L. Di Gennaro, MD, Assistant Professor, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 24849 Academic Enrichment Fund
Record Dates: First submitted 2013-05-02; First posted 2013-05-07 (Estimated); Results first posted 2020-08-13 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Agitation
Keywords: acupuncture; pediatric; critical care; mechanical ventilation; sedation; comfort
MeSH Terms: conditions — Psychomotor Agitation | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acupuncture (Experimental): Acupuncture treatment three times per week for up to two weeks.
  Interventions: Device: acupuncture
- Sham Acupuncture (Sham Comparator): Sham acupuncture three times per week for up to two weeks
  Interventions: Device: sham acupuncture

INTERVENTIONS:
Device: acupuncture — Patients randomized to active treatment will receive acupuncture treatment with press needles (small acupuncture needles manufactured with attached bandage that makes the needle flush with skin) at sites GV 24.5 or GV20, Ht 7 or Ht 3, Ki 3, Lr 3, LI 4 or LI 11, Lu 7 or Lu 5, Sp6, ST 36, using up to 15 points per patient three days per week for the duration of mechanical ventilation (maximum of 14 calendar days from the time of the first acupuncture treatment). We will also apply a seed magnet at ear shen men position for 4 hours on treatment days.
  Other Names: Pyonex Singles, Seirin® (0.20 mm diameter, 1.5 mm long)
  Arms: Acupuncture
Device: sham acupuncture — Patients randomized to sham treatment will receive sham acupuncture with similarly appearing bandages placed without press needles attached at sites GV 24.5 or GV20, Ht 7 or Ht 3, Ki 3, Lr 3, LI 4 or LI 11, Lu 7 or Lu 5, Sp6, ST 36, using up to 15 points per patient three days per week for the duration of mechanical ventilation (maximum of 14 calendar days from the time of the first acupuncture treatment). We will also apply a similarly appearing bandage without seed magnet underneath at ear shen men position for 4 hours on treatment days.
  Other Names: Pyonex Singles, Seirin® (bandage only, no needle)
  Arms: Sham Acupuncture

SUMMARY:
The purpose of this study is to determine whether acupuncture is effective at improving comfort in children on a ventilator in the intensive care unit. Our hypothesis is that the patients receiving acupuncture will require less medications to keep them comfortable than those who receive sham or fake acupuncture.

DETAILED DESCRIPTION:
Rationale: Use of narcotics and benzodiazepines is common in the pediatric intensive care unit (PICU) to alleviate pain and anxiety, especially for patients who are mechanically ventilated. Pain control and sedation decrease oxygen consumption, facilitate mechanical ventilation, ensure patient safety and help patients tolerate nursing care. However, these medications can also have negative consequences. Patients receiving greater amounts of pharmacologic sedation in the intensive care unit (ICU) have longer duration of mechanical ventilation and ICU length of stay. In fact, daily interruption of sedation shortens duration of mechanical ventilation and ICU length of stay. Sedatives have also been associated with development of delirium in ICU patients and linked to delusional and disturbing memories and post-traumatic stress disorder (PTSD) after recovery from critical illness. Benzodiazepines and opiates are associated with abnormal sleep architecture. Furthermore, patients experience tolerance, physical dependency and withdrawal from these agents. Lastly, there is evidence that sedatives, anesthetics and opiates are associated with neurotoxicity in animal studies leading to growing concern about the potential effects of these agents on the developing brains of children.

Novel Approach: In light of these negative aspects of pharmacologic sedation, we are looking for alternative ways to provide comfort to critically ill children in the PICU. Acupuncture has been found to be effective in reducing anxiety, acute pain, procedural pain, post-operative pain, chronic pain, headache, infant colic, and has been found to reduce anesthetic requirement during surgery.

Study Plan: We plan to randomize patients 6 months - 17 yrs old who are receiving mechanical ventilation in the PICU to either acupuncture or sham acupuncture as an adjunct to standard of care pharmacologic sedation as prescribed by the PICU medical team caring for the patients. Our hypothesis is that those patients receiving acupuncture will require less medications to keep them comfortable. Our study is powered (80%) to detect a 33% decrease in pharmacologic sedation/analgesia.

ELIGIBILITY:
Inclusion Criteria:

* age ≥6 months to <18 years
* intubated and mechanically ventilated
* patient requires pharmacologic sedation/analgesia to tolerate mechanical ventilation
* ≤72 hours of mechanical ventilation at time of enrollment with anticipated need of mechanical ventilation for at least ≥48 hours more (in order to be able to receive at least one acupuncture session)
* approval of treating physician

Exclusion Criteria:

* underlying neurologic condition that could impact sedation/analgesia needs
* coagulopathy (inr ≥ 1.8) or history of spontaneous bruising
* thrombocytopenia (platelets <20,000 that has not been treated with a platelet transfusion)
* hemodynamic instability (on continuous infusion of vasopressor or inotrope)
* sepsis or bacteremia on antibiotic therapy <24 hours
* severe generalized skin disorder (e.g., epidermolysis bullosa, Stevens-Johnson)
* ward of state
* being treated with therapeutic level of systemic anticoagulation (e.g., heparin with unfractionated heparin activity level ≥0.3, enoxaparin with low molecular weight heparin activity level ≥0.5, warfarin with inr ≥1.8)
* immunosuppressed (on chemotherapy {e.g., daunorubicin, vincristine}, immunosuppressive medications {e.g., sirolimus, tacrolimus, cyclosporine, mycophenolate mofetil, high dose steroids >4mg/kg/day}, or immunosuppressive biologics {e.g., thymoglobulin, etanercept, infliximab, adalimumab, rituximab})

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2013-03; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jane L Di Gennaro, MD, MS, Principal Investigator — Seattle Children's Hopsital; Anne Lynn, MD, Principal Investigator — Seattle Children's Hospital
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States

REFERENCES:
- [Derived] Kudchadkar SR, Berger J, Patel R, Barnes S, Twose C, Walker T, Mitchell R, Song J, Anton B, Punjabi NM. Non-pharmacological interventions for sleep promotion in hospitalized children. Cochrane Database Syst Rev. 2022 Jun 15;6(6):CD012908. doi: 10.1002/14651858.CD012908.pub2. PMID 35703367

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Acupuncture | Sham Acupuncture
Started | 10 | 7
Completed | 10 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acupuncture | Sham Acupuncture | Total
Number analyzed (Participants) | 10 | 7 | 17
Age, Continuous [Median (Full Range); unit: years] | 2.4 [0.7 to 16.8] | 1.0 [0.8 to 3.6] | 1.7 [0.7 to 16.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 5 | 2 | 7
Region of Enrollment [Number; unit: participants]
  United States | 10 | 7 | 17
PRISM III [Median (Full Range); unit: units on a scale] — Pediatric Risk of Mortality III score: Physiology based illness severity score for critically ill children in the pediatric intensive care unit. The total score ranges from 0 to 74, with higher score associated with worse prognosis.
  units on a scale | 0 [0 to 3] | 3 [0 to 14] | 0 [0 to 14]

OUTCOME MEASURES:

1. Primary Outcome: Average Daily Dexmedetomidine mcg/kg/Day
Description: Measured total amount of dexmedetomidine received from time of first acupuncture or sham treatment to extubation, normalized per weight and time on study (1st study treatment to extubation).
Time Frame: from time of first acupuncture/sham treatment till time of extubation
Measure: Mean (Standard Deviation); unit: mcg/kg/day
Arm/Group | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 10 | 7
mcg/kg/day | 11.08 (9.37) | 17.42 (6.36)

2. Primary Outcome: Average Daily Morphine Equivalents (mg/kg/Day)
Description: Measured total amount of morphine equivalent received from time of first acupuncture or sham treatment to extubation, normalized per weight and time on study (1st study treatment to extubation).
Time Frame: from time of first acupuncture/sham treatment till time of extubation
Measure: Mean (Standard Deviation); unit: mg/kg/day
Arm/Group | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 10 | 7
mg/kg/day | 1.04 (0.68) | 1.61 (1.12)

3. Primary Outcome: Average Daily Midazolam Equivalents (mg/kg/Day)
Description: Measured total amount of midazolam equivalent received from time of first acupuncture or sham treatment to extubation, normalized per weight and time on study (1st study treatment to extubation).
Time Frame: from time of first acupuncture/sham treatment till time of extubation
Measure: Mean (Standard Deviation); unit: mg/kg/day
Arm/Group | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 10 | 7
mg/kg/day | 0.73 (1.03) | 0.97 (0.80)

4. Primary Outcome: Average Daily Sedation Score
Description: To capture a global view of sedation and account for the combination of medications received, we also calculated an average daily 'sedation score' normalized for weight from the time of first treatment through extubation. The sedation score is a summary measure of sedative and analgesic exposure for mechanically ventilated children in the ICU. This score incorporates opioids, benzodiazepines, barbiturates, chloral hydrate, propofol, and antihistamines. Morphine and midazolam equivalents of 0.1 mg/kg, pentobarbital 2 mg/kg, chloral hydrate 50 mg/kg, any propofol use, and any phenobarbitol use are each allocated one point, while any antihistamine use receives a score of 0.5 (Randolph 2002, Curley 2005). We modified this score to include dexmedetomidine, assigning 1 point for 1 μg/kg of dexmedetomidine. The minimum value possible is zero, and there is no pre-defined maximum value. A higher score indicates higher dose of sedation medications (normalized by weight).
Time Frame: from time of first acupuncture/sham treatment till time of extubation
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 10 | 7
score on a scale | 29.0 (20.8) | 43.4 (18.4)

5. Secondary Outcome: Number of Participants With Skin Ulceration at Acupuncture/Sham Sites
Time Frame: From time of first treatment through 2 to 3 days after last treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 10 | 7
Participants | 0 | 0

6. Secondary Outcome: Number of Participants With Hematoma at Acupuncture/Sham Sites
Time Frame: From time of first treatment through 2 to 3 days after last treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 10 | 7
Participants | 0 | 0

7. Secondary Outcome: Number of Participants With Cellulitis at Acupuncture/Sham Sites
Time Frame: From time of first treatment through 2 to 3 days after last treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 10 | 7
Participants | 0 | 0

8. Secondary Outcome: Number of Participants Who Are Diagnosed With Bacteremia During the Study
Time Frame: From time of first treatment through 2 to 3 days after last treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 10 | 7
Participants | 0 | 0

9. Secondary Outcome: Number of Participants Who Are Diagnosed With Septic Shock During the Study
Time Frame: From time of first treatment through 2 to 3 days after last treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 10 | 7
Participants | 0 | 0

10. Secondary Outcome: Death While Enrolled in Study
Time Frame: From time of first treatment through 2 to 3 days after last treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 10 | 7
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: From time of first treatment through 2 to 3 days after last treatment.
Description: Adverse events will be identified through review of the patient's hospital chart, discussion with treating medical team, and physical examination (to assess skin findings) every Monday, Wednesday and Friday while enrolled in the active phase of the trial (receiving acupuncture or placebo) and one additional evaluation 2 to 3 days after completing the last session of acupuncture or placebo (the Monday, Wednesday or Friday following the last study treatment).
Arm/Group | Acupuncture | Sham Acupuncture
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/7
Other Adverse Events (participants affected / at risk) | 0/10 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No